CLINICAL TRIAL: NCT02133209
Title: MRI Outcomes of Mindfulness Meditation for Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00091884; R01AT007176 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-05-07 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Migraine
Keywords: migraine; headache; meditation; mindfulness based stress reduction; MBSR
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stress Management for Headaches (Active Comparator): This intervention involves a standardized stress management for headaches (SMH) group intervention that focuses on stress and general stress management skills for managing migraine headaches.
  Interventions: Behavioral: Stress Management for Headaches
- Mindfulness Based Stress Reduction (Active Comparator): Intervention involves a standardized mindfulness-based stress reduction (MBSR) group intervention following the guidelines originally conceived and developed by the Center for Mindfulness in Medicine, Health Care and Society at the University of Massachusetts. The intervention also included an extended period of training in addition to the usual 8 weeks.
  Interventions: Behavioral: Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Mindfulness Based Stress Reduction (MBSR) involves focused attention while practicing moment-to-moment nonjudgmental awareness of the self with the goal of achieving emotional balance and clarity of thought. There will be 8 weekly sessions and a half day retreat followed by 4 bi-weekly sessions over a period of 4 months.
  Arms: Mindfulness Based Stress Reduction
Behavioral: Stress Management for Headaches — Intervention involves a standardized stress management for headaches (SMH) group intervention that focuses on stress and general stress management skills, headache symptoms and their management, sleep hygiene, and healthy eating. There will be 8 weekly sessions followed by 4 bi-weekly sessions over a period of 4 months.
  Arms: Stress Management for Headaches

SUMMARY:
112 migraine subjects will be initially randomly assigned to Mindfulness-Based Stress Reduction (MBSR) or a Stress Management for Headache group (SMH). Outcomes, including headache frequency and impact and brain activity, will be assessed at baseline, prior to intervention, and at 3-, 6-, and 12-months.

DETAILED DESCRIPTION:
Subjects in the MBSR group undergo a standardized 8-week MBSR course plus an additional 4 sessions over another 8 weeks that further emphasize and train subjects on MBSR concepts and skills. The SMH group will have 12 sessions spread out in a similar fashion to MBSR. Clinical outcomes are compared between groups at 3, 6, and 12 months to assess efficacy of MBSR. MRI scans are performed at baseline, 3 months, and 6 months changes in MRI metrics after MBSR and changes in MRI metrics associated with long-term MBSR practice. 30 healthy controls will also undergo MRI scanning to determine abnormal brain activity and structure in migraineurs compared to healthy controls across the 6 month period of observation.

ELIGIBILITY:
Inclusion Criteria

* Are between 18 and 65 years of age
* Report between 4 and 14 headaches over 28 days
* Have a history of migraines lasting at least 1 year
* Are not currently using opioid ("narcotic") pain medication

Exclusion Criteria

* Are unable to undergo MRI
* Pregnant, lactating, or planning to become pregnant
* Current use of opioid medications

Inclusion Criteria for Healthy Volunteers (same exclusion criteria)

* Are between 18 and 65 years of age
* Free of any acute or chronic pain condition and reports no history of migraines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in headache frequency and impact | Baseline, 3, 6, and 12 months
  Headache days per 28 days and headache-related disability (HIT-6)
Change in gray matter volume | Baseline, 3, and 6 months
  Gray matter volume in the insula, dorsolateral prefrontal cortex, and cingulate
Change in Brain Function | Baseline, 3, and 6 months
  Overall activation of the dorsolateral prefrontal cortex and the task-positive cognitive network, and resting state connectivity to the insula

SECONDARY OUTCOMES:
Change in headache intensity | Baseline, 3, 6, and 12 months
  Change in headache intensity
Change in Brain Structure | Baseline, 3, and 6 months
  Gray matter volume and white matter tracts across the whole brain
Change in Whole Brain Function | Baseline, 3, and 6 months
  Cognitive-related activity, pain-related activity, and resting state across the whole brain

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Haythornthwaite, Ph.D., Study Director — Johns Hopkins University; David Seminowicz, Ph.D., Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - University of Maryland School of Dentistry, Baltimore, Maryland
  - Johns Hopkins University, Bayview Medical Campus, Baltimore, Maryland

REFERENCES:
- [Derived] Burrowes SAB, Goloubeva O, Keaser ML, Haythornthwaite JA, Seminowicz DA. Differences in gray matter volume in episodic migraine patients with and without prior diagnosis or clinical care: a cross-sectional study. J Headache Pain. 2021 Oct 23;22(1):127. doi: 10.1186/s10194-021-01340-5. PMID 34688253
- [Derived] Burrowes SAB, Goloubeva O, Stafford K, McArdle PF, Goyal M, Peterlin BL, Haythornthwaite JA, Seminowicz DA. Enhanced mindfulness-based stress reduction in episodic migraine-effects on sleep quality, anxiety, stress, and depression: a secondary analysis of a randomized clinical trial. Pain. 2022 Mar 1;163(3):436-444. doi: 10.1097/j.pain.0000000000002372. PMID 34407032